CLINICAL TRIAL: NCT00458536
Title: Vaccination of Patients With Renal Cell Cancer With Dendritic Cell Tumor Fusions and GM-CSF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, David Avigan, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-117
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Renal Cancer
Keywords: GM-CSF; vaccine; debulking nephrectomy; dendritic cells
MeSH Terms: conditions — Kidney Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Patients treated with DC/RCC vaccine to evaluate for treatment-limiting toxicity
  Interventions: Biological: Dendritic Cell Tumor Fusion Vaccine; Drug: Granulocyte Macrophage Colony Stimulating Factor (GM-CSF)
- Cohort 2 (Experimental): Patients treated with DC/RCC vaccine to evaluate response
  Interventions: Biological: Dendritic Cell Tumor Fusion Vaccine; Drug: Granulocyte Macrophage Colony Stimulating Factor (GM-CSF)

INTERVENTIONS:
Biological: Dendritic Cell Tumor Fusion Vaccine — 3 vaccinations at three week intervals
Drug: Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) — Combined with the vaccine in the remaining subjects after the first 6 are enrolled.

SUMMARY:
The main purpose of this study is to test the safety of the dendritic cell/tumor fusion study vaccine in combination with a laboratory-made agent called Granulocyte Macrophage Colony Stimulating Factor (GM-CSF). Another purpose is to determine the type and severity of any side effects associated with this study vaccine. GM-CSF is similar to a substance in the body that stimulates the production of white blood cells. To create the study vaccine, cells will be removed from the participants tumor and fused with dendritic cells which are obtained from the participants blood. Dendritic cells are responsible for immune responses to "foreign" substances that enter the body. Animal studies have shown that these fused cells can stimulate powerful anti-tumor responses.

DETAILED DESCRIPTION:
* Patients are being asked to participate if they have chosen to undergo a "debulking nephrectomy" (surgery to remove a tumor of the kidney, but not all of the cancer cells in their body) as a standard treatment for kidney cancer or they have tumor lesions that are accessible and are being removed to treat or diagnose their cancer.
* Participants enrolled in this study will be assigned to receive a particular dose of the dendritic cell/tumor fusion vaccine cells. The dose will be determined by when they are enrolled in the study. There are two cohorts to this study. The first cohort will be given the vaccine alone. If the vaccine is well tolerated then we will proceed to the second cohort. The second cohort will receive GM-CSF in addition to the vaccine.
* Tumor cells will be collected to make the study vaccine. Based on the location of the cancer, a decision will be made as to the best approach to obtain these cells.
* Participants will undergo a procedure known as leukapheresis in order to obtain their dendritic cells. Prior to this procedure they will receive 1 to 2 injection of GM-CSF to help increase their white blood cell count.
* If sufficient numbers of cells are obtained, tumor cells and dendritic cells will be fused (mixed) together in the laboratory and divided into the appropriate doses for administration.
* The treatment will consist of 3 vaccinations of fused cells given by an injection under your skin at 3-week intervals. The first six participants will receive only the study vaccine. The remaining participants will receive the study vaccine combined with GM-CSF.
* If enough vaccine cannot be made for the participant to receive 3 doses, the participant may receive only 2 doses of the study vaccine.
* Approximately 3 to 4 tablespoons of blood will be collected at certain times for testing the immune system and to determine if the study vaccine has increased the immune response against the tumor cells. Weekly visits for physical exam, assessment of adverse events and safety labs will be conducted.
* Regular blood draws will be done for at least 6 months following the completion of the study to follow safety labs and to monitor the immune response. Monthly physical exams will be performed following the last injection of the study vaccine. At one month, three months, and six months following the date the participant received the last study vaccine, they will have a CT scan to see if the study vaccine has affected their disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IV renal cancer who have not received prior chemotherapy or biological therapy
* Patients who are to undergo debulking nephrectomy for independent clinical indications or patients with other sites of accessible disease
* Tumor tissue should be at least 2.0cm in longest dimension
* Patients should meet prognostic criteria for intermediate or favorable risk disease as defined by Motzer criteria
* Measurable metastatic disease as defined by a lesion of at least 1cm outside the lesion used for vaccine generation and exclusive of bony metastases
* ECOG Performance Status of 0-2 with greater than six week life expectancy
* 18 years of age or older
* Lab results within range outlined in protocol

Exclusion Criteria:

* Patients who have received prior chemotherapy
* Clinical evidence of CNS disease. Patients with a history of treated brain metastasis must be stable with no evidence of disease for 3 months
* HIV positive
* Serious intercurrent illness such as infection requiring IV antibiotics, or significant cardiac disease characterized by significant arrhythmia, unstable ischemic coronary disease or congestive heart failure
* Pregnant of lactating women
* History of clinically significant venous thromboembolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-10; Primary Completion 2014-12 (Actual); Study Completion 2023-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Treated With Vaccine: Patients with renal cell carcinoma following debulking nephrectomy who receive at least 2 doses of DC/renal fusion vaccine.
Period: Overall Study
Arm/Group | Patients Treated With Vaccine
Started | 38
Completed | 19
Not Completed | 19
Not completed — Disease progression prior to treatment | 7
Not completed — Unable to make vaccine | 3
Not completed — No measurable disease after surgery | 2
Not completed — Did not have renal cell carcinoma | 2
Not completed — Patient did not have surgery | 1
Not completed — Ineligible due to toxicity | 1
Not completed — Withdrawal by Subject | 1
Not completed — Progressive disease during treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Patients Treated With Vaccine
Number analyzed (Participants) | 19
Age, Customized [Median (Full Range); unit: years] | 56 [43 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Associated With Vaccination With Mature DC/Tumor Fusion and GM-CSF
Time Frame: 5 years
Population: Adverse events potentially related to vaccination were largely restricted to injection site reactions. 12 of the 19 patients experienced vaccine site reactions.
Measure: Number; unit: participants
Arm/Group | Patients Treated With Vaccine
Number analyzed (Participants) | 19
participants | 12

2. Secondary Outcome: To Determine if Cellular and Humoral Immunity is Induced by Serial Vaccination With DC/Tumor Fusion Cells and GM-CSF
Time Frame: 5 years
Reporting Status: Not Posted

3. Secondary Outcome: to Correlate Immunologic Response Following Vaccination.
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs were collected over the course of the study while patients were being treated. This spanned 4 years.
Arm/Group | Patients Treated With Vaccine
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 16/19
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With Vaccine (N=19)
Injection Site Reaction (Investigations) | 12 (25)
Bruising (at site of vaccine) (Blood and lymphatic system disorders) | 3 (7)
Arthralgias (Musculoskeletal and connective tissue disorders) | 1 (2)
Urticaria (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No